CLINICAL TRIAL: NCT06659939
Title: Method for bAdge-dosi Monitoring of X-ray Exposure Values in Operating Theatre Surgery: a Multicentre Randomised Trial
Brief Title: Method for bAdge-dosi Monitoring of X-ray Exposure Values in Operating Theatre Surgery
Acronym: MAVERIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR240215 - MAVERIC
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: X-Ray
Keywords: radioprotection; dosimeter; surgical staff; operating room; radiation monitoring; Badge

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- TEST group: The TEST group's participants will be randomized in order to either wear the dosimeter alone (as usual) or the dosimeter associated with the access badge of the hospital "badge-dosi".
  The participants are working in the operating room and are exposed to X-rays
- LIFE group: The LIFE group participants will wear a dosimeter associated with the access badge of the hospital "badge-dosi".
  The participants are working in the same hospital as the TEST group, but they are not exposed to any radiation at work.
- HOME group: The HOME group participants will have a dosimeter alone which will be stored at home. The participants are working in the same hospital as the TEST group.

SUMMARY:
Surgical procedures involving X-rays in the operating room have increased in recent years, thereby increasing the exposure of operating room staff to ionizing radiation. An individual dosimeter makes it possible to record the radiation exposure to which these personnel are exposed. However, it has been noticed that these dosimeters are not thoroughly worn, consequently the radiation doses recorded are not reliable.

In order to increase the proportion of dosimeters systematically worn in the operating room, we study the impact of the association of the passive dosimeter with the hospital access badge (forming the Badge-Dosi). A first pilot study was carried out at Tours University Hospital showing the effectiveness of this concept. With the present study, we carry out a multicenter study. Our hypothesis is that the Badge-Dosi allows a significant increase of dosimeter use in the operating room, which improves the reliability of the monitoring of personnel.

ELIGIBILITY:
Inclusion Criteria:

TEST group :

* People working in the operating room at least 80% of the time (excluding people working less than 80% of the time).
* Have been monitored by a delayed-reading dosimeter for at least 1 year.
* Carry an access card (i.e. be the holder).

LIFE group :

* Person working in the same centre as the people in the TEST group.
* Person not exposed to radiation at their workstation
* Holder of an access card

HOME group :

- Person working in the same centre as people in the TEST Group and live near the center

Exclusion Criteria:

For all Groups :

* Person objecting to data processing
* Interns/externs/non-permanent staff likely to change jobs during the study period
* Person who had a nuclear medicine examination within 15 days before the start of the study
* Anyone who had internal vectorised therapy with iodine-131 or Lu-177 within 30 days before the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: staff exposed to X-rays working in the operating room (TEST group)
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Improve the wearing of dosimeters by staff exposed to X-rays and working in the operating room thanks to the BadgeDosi solution in order to make the exposure measurements taken more reliable and interpretable compared to the passive dosimeter alone. (TES | 6 months
  Passive dosimeter wearing status (alone versus BadgeDosi) assessed once by an independent observer over the M6 period (during the sixth month of the study, TEST group).

SECONDARY OUTCOMES:
Evaluate the wearing rate the passive dosimeter assessed by questionnaire at M0, M3 and M6 (TEST group) | Month 0, month 3 and month 6
  Passive dosimeter wearing rate is assessed at M0, M3 and M6 by a declarative questionnaire (TEST group).
Study the evolution of radiation read on the BadgeDosi versus passive dosimeter alone among agents working in the operating room (TEST group). | Month 3 and month 6
  Difference in radiation measured in mSv between the BadgeDosi and the dosimeter alone (TEST group, M3 and M6).
Study the variations of doses of a control group wearing the BadgeDosi but not exposed to ionizing radiation as part of their activity in the hospital (VIE group). | Month 3 and month 6
  Difference in radiation measured in mSv between the dosimeters of the TEST group and of the VIE control group (M3 and M6).
Collect user feedback on the ergonomics the BadgeDosi (TEST and VIE groups). | Month 3 and month 6
  Questionnaire on feedback (ergonomics, usability, satisfaction) from the TEST group and the VIE control group (M3 and M6).
Monitor natural radioactivity between the healthcare center and the staff's homes. Special care is taken so the distribution of the places of residence of the staff around the hospital is represented (HOME group). | Month 3 and month 6
  Difference in radiation measured in mSv between healthcare center and staff's homes (HOME control group, M3 and M6).
Collect user feedback on the use of the UV box placed in the changing rooms for disinfection of personal objects (including but not limited to the BadgeDosi) entering the OR department (TEST groups). | Month 3 and month 6.
  Questionnaire on feedback from the TEST group M3 and M6

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - University hospital, Orléans
  - University hospital, Toulouse
  - University hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided